CLINICAL TRIAL: NCT05567913
Title: Change in Perceived Stress Level and Stress-related Symptoms in Elementary School Students During Active Stress Prevention Work With the Addition of a Physiotherapist to the School's Student Health Team.
Brief Title: Change i Perceived Stress in School-age Students When Adding Physiotherapists to a School's Health Team.
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Dals-Ed Municipality (Unknown)
Responsible Party: Principal Investigator, Anna Bergenheim, RPT, PhD, Vastra Gotaland Region
Other Study IDs: VGFOUFBD976982
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stress-related Problem
Keywords: School health services; Physical therapy modalities; Mental health; Child; Adolescent
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
School stress and performance requirements have been shown to contribute to mental illness among children and young people.

Student health teams have an important role regarding mental health of children and young people. Swedish student health teams include various health and pedagogical professionals, but physiotherapists are uncommon, despite the good effects school-related physical activity interventions have had on reducing anxiety and improving well-being in children and young people.

Haga School, Dals-Ed has now employed physiotherapists as part of the student health team to support students in learning to define, reduce and manage stress.

The purpose of the research project is to investigate changes in perceived stress level and stress-related symptoms, as well as study results and absence from school during two years for students in grades 4 to 9 at Haga School. A questionnaire will be sent out on four occasions over two years. Group level statistics on study results and school absence will be compared with years previous to the introduction of the school physiotherapist. The research contributes to increased knowledge about effects of having a physiotherapist as part of a student health team in Sweden.

DETAILED DESCRIPTION:
School stress and performance requirements have been shown to contribute to mental illness among children and young people.

Student health teams have an important role regarding mental health of children and young people. Swedish student health teams include various health and pedagogical professionals, but physiotherapists are uncommon, despite the good effects school-related physical activity interventions have had on reducing anxiety and improving well-being in children and young people.

Haga School, Dals-Ed has now employed physiotherapists as part of the student health team to support students in learning to define, reduce and manage stress.

The purpose of the research project is to investigate changes in perceived stress level and stress-related symptoms, as well as study results and absence from school during two years for students in grades 4 to 9 at Haga School. A questionnaire will be sent out on four occasions over two years. Group level statistics on study results and school absence will be compared with years previous to the introduction of the school physiotherapist. The research contributes to increased knowledge about effects of having a physiotherapist as part of a student health team in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Registered students in grades 4-9 at Haga School in Dals-Ed, Sweden

Exclusion Criteria:

* None

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All registered students in grade 4-9 at Haga school Dals-Ed, Sweden 2022-2025.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Measured with single question on questionnaire with 4 possible levels to choose from, ranging from "not at all" to "very much".
Reasons for stress | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question about stressors chosen from a list of 7 stressors or no stressors
School stress factors School stress factors School stress factors | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question about factors that contribute to perceived stress in school, chosen from a list of 16 stressors.

SECONDARY OUTCOMES:
Stress-related symptoms | Change between inclusion and 8 month, 12 and 20 month follow-ups
  Measured with number of stress-related symptoms chosen from a list of 7 symptoms or no symptoms.
Prevalence of specific stress-related symptoms | Change between inclusion and 8 month, 12 and 20 month follow-ups
  Number of students who report each specific symptom from a list of 7 symptoms or no symptoms.
Stress-alleviating factors | Change between inclusion and 8 month, 12 and 20 month follow-ups
  Single question regarding handling of stress symptoms, chosen from list of 9 suggestions or open-ended answer.
Headache prevalence | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question regarding prevalence of headache during the last month with 5 possible levels, ranging from "never" to "always".
Stomach-ache prevalence | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question regarding prevalence of stomach-ache during the last month with 5 possible levels, ranging from "never" to "always".
Prevalence of irritability | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question regarding irritation or bad mood during the last month with 5 possible levels ranging from "never" to "always".
Prevalence of depressive feelings | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question regarding feeling sad or depressed feelings during the last month with 5 possible levels ranging from "never" to "always".
Sleeping habits | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question about sleep quality with 5 possible answers ranging from "very bad" to "very good".
Well-being at school | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question regarding well-being at school with 5 possible levels, ranging from "very bad" to "very good".
Physical activity | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question about amount of physical activity during the last 7 days, with 8 possible levels, ranging from "less than 1 hour" to "more than 10 hours"
Transportation to school | Change between inclusion and 8 month, 12 and 20 month follow-ups.
  Single question about commuting to school with four possible answers, walking, bicycling, bus, car/moped.
School absence | Change between school-year 2021-2022 and 2023-2024.
  Group level school absence retrieved from school statistics. Measured in number of days. days.
Study results | Change between school-year 2021-2022 and 2023-2024.
  Group level study results for each grade. Measured in grades E-A.
Eligibility upper-level secondary school | Change between school-year 2021-2022 and 2023-2024.
  Group level eligibility for upper-level secondary school programs for students in Grade 9. Measured in number of students eligible for upper-level secondary school.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bergenheim, PhD, Principal Investigator — Region Västra Götaland, University of Gothenburg
Locations (1):
- Haga School, Ed, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers than the participating research group.